CLINICAL TRIAL: NCT00340418
Title: Mechanisms of Lung Allograft Rejection
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905182; 05-E-N182
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-04-13

CONDITIONS: Lung Transplant; Chronic Allograft Rejection
Keywords: Bronchoalveolar Lavage; Acute Rejection; Chronic Rejection; Genetic Polymorphisms; Innate Immunity; Lung Transplantation; Lung Allograft Rejection

SUMMARY:
This study will explore the ways in which lung transplants are rejected. A series of experiments will evaluate the differences in airway gene expression. Lung transplantation has become an important option for patients with advanced lung disease. More than 10,000 patients have received them to date, and about 1,200 transplant operations are performed worldwide each year. Although short-term survival has continued to improve, the 5-year survival rate is less than 50%. Most posttransplant deaths are directly or directly caused by chronic lung rejection, a condition of scarring that worsens lung function. .

Patients ages 18 and older who have received lung transplants, who are undergoing bronchoscopy as part of the usual care after transplant, and who are not pregnant may be eligible for this study.

Bronchoscopy and other procedures performed during this study are done only by doctors with special training. They will take a total of 30 to 60 minutes. During a bronchoscopy, patients will lie on a flat bed. They will be awake and follow instructions. First they will breathe Xylocaine (lidocaine), an anesthetic mist, for 8 to 10 minutes. That will lessen the discomfort of a small flexible tube called a bronchoscope that will be guided through the back of the patient's mouth or nose and into the breathing tubes. When the flexible tube is placed, patients will not be able to speak. They will receive the medication Versed (midazolam), to make them relaxed and not remember most of the procedure, and fentanyl, to decrease the possibility of feeling pain. These medications will be given through a narrow tube feeding into a small needle placed into a vein in the arm. The risks of the tube placed in the vein include bleeding, swelling, redness, and pain. Side effects from the medications may include stomach upset, heart palpitations (awareness of heartbeat), and changes in blood pressure. Patients will be carefully monitored for heart rate, blood pressure, breathing, and oxygen levels.

During the bronchoscopy, a procedure called bronchoalveolar lavage is done, in which a small amount of germ-free salt water is injected into through the bronchoscope into the lung and immediately suctioned back, thus washing the lining of the airways and checking for infection and rejection of the transplanted lungs. About 1 or 2 tablespoons of fluid will be collected for analysis. Also, an endobronchial brush biopsy may be performed. A small brush removes some of the cells from the surface of the airway. These cells will be sent to a laboratory at Duke University Health system to analyze the signals from the cells that may eventually led to scarring and chronic rejection of the lungs. Then, an endobronchial forceps biopsy is performed, in which one or two small pieces, each about the size of a grain of rice, of the lining of the lung's large airways is removed. A small surgical tool like tweezers is passed into the lung. Risks of biopsies may include bleeding, injury to the lung, or an air leak in the lung.

This study will not have a direct benefit for participants. However, it is hoped that information gathered will enhance researchers' understanding of how lung rejection occurs.

DETAILED DESCRIPTION:
Lung transplantation has emerged as a viable therapeutic option in the care of patients with advanced pulmonary parenchymal and pulmonary vascular disease. Currently, over 10,000 patients have received lung transplantation with approximately 1200 transplant operations performed worldwide each year. Short term survival after lung transplantation has continued to improve since the widespread application of this procedure and one-year survival at most centers now approaches 80%. Unfortunately, long-term outcomes after lung transplantation are disappointing with five-year survival below 50%. Most posttransplant deaths are due directly or indirectly to the development of chronic allograft rejection, which affects approximately 50% of all five-year survivors. Acute rejection is the major risk factor for the development of chronic rejection. Chronic lung rejection leads to a condition of irreversible fibrosis and obliteration of the small to medium size bronchioles known as obliterative bronchiolitis (OB). Very little is known about the pathogenic mechanisms that lead to the development of OB. Furthermore, it is unclear why acute rejection leads to the development of chronic rejection in some but not all patients. In order to better understand the mechanisms of OB we propose a series of experiments designed to evaluate differences in airway gene expression in a series of lung transplant recipients with and without acute rejection.

ELIGIBILITY:
* INCLUSION CRITERIA:

All adult (18 and older) lung transplant recipients who are undergoing bronchoscopy as part of the usual posttransplant care will be eligible.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2005-06-23; Study Completion 2007-04-13

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - NIEHS, Research Triangle Park, Research Triangle Park, North Carolina

REFERENCES:
- [Background] Tazelaar HD, Yousem SA. The pathology of combined heart-lung transplantation: an autopsy study. Hum Pathol. 1988 Dec;19(12):1403-16. doi: 10.1016/s0046-8177(88)80233-8. PMID 3142814